CLINICAL TRIAL: NCT04109534
Title: Investigation of the Effect of a Dietary Fatty Acid Supplementation on Symptoms and Bronchial Inflammation in Patients With Asthma and House Dust Mite Allergy After Repeated Allergen Challenge
Brief Title: Effect of a Dietary Fatty Acid Supplementation on Symptoms and Bronchial Inflammation in Patients With Asthma
Acronym: LCPUFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stefan Zielen (Other)
Responsible Party: Sponsor-Investigator, Stefan Zielen, Professor, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-263
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Allergic Asthma; Allergy to House Dust Mite
Keywords: allergic asthma,; house dust mite allergy; bronchial allergen provocation; LCPUFAs
MeSH Terms: conditions — Dust Mite Allergy | interventions — Bronchial Provocation Tests; Nasal Provocation Tests

STUDY DESIGN:
Intervention Model Description: Placebo-controlled prospective study
Who Masked: Participant, Investigator
Masking Description: LCPUVAS and Placebo are provided in sealed bags
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo comparator 20 patients aged 18-45 years with a diagnosis of HDM induced allergic asthma and an increase of exhaled NO of 30% after BAP will be randomized to the Placebo Comparator
  Interventions: Diagnostic Test: Bronchial allergen provocation (BAP); Diagnostic Test: Nasal provocation test (NPT); Diagnostic Test: Methacholine test; Diagnostic Test: Peak nasal expiratory flow (PNIF)
- Verum (Active Comparator): PUFAS: 2640 mg of middle-chain and polyunsaturated fatty acids 20 patients aged 18-45 years with a diagnosis of HDM induced allergic asthma and an increase of exhaled NO of 30% after BAP will be randomized to the Active Comparator
  Interventions: Diagnostic Test: Bronchial allergen provocation (BAP); Diagnostic Test: Nasal provocation test (NPT); Diagnostic Test: Methacholine test; Diagnostic Test: Peak nasal expiratory flow (PNIF)

INTERVENTIONS:
Diagnostic Test: Bronchial allergen provocation (BAP) — Nebulized Dermatophagoides farina administered at following doses: 10AE, 20 AE, 40 AE, 80 160 AE, etc… until the FEV1 decreases 20% below the initial FEV1-value
Diagnostic Test: Nasal provocation test (NPT) — Dermatophagoides farina will be administered in both nostrils
Diagnostic Test: Methacholine test — Nebulized metacholine will be administered at following doses: 0,01mg, 0,1mg, 0,4mg, 0,8mg und 1,6mg until the FEV1 decreases 20% below the initial FEV1-value
Diagnostic Test: Peak nasal expiratory flow (PNIF) — Comparison of peak nasal expiratory flow (PNIF) after NPT between groups

SUMMARY:
The proposed study will investigate the effect of a polyunsaturated fatty acid / lipid mixture (LCPUFAs) on the clinical symptoms, bronchial inflammation and lung function in allergic asthma in a bronchial allergen provocation (BAP) model. For this purpose, patients with stable episodic asthma and dust mite allergy will underwent BAP before and after supplementation with LCPUFAs. The clinical symptoms, bronchial inflammation, exhaled NO increase and lung function decline (FEV1) will be analyzed.

DETAILED DESCRIPTION:
Asthma is a chronic lung disease, which is characterized by recurrent obstruction, a hypersensitivity and a chronic inflammation of the airway. It is known that LCPUVAs could reduce the production of inflammatory mediators. In addition, LCPUVAs can improve pulmonary function, with a concurrent reduction in bronchodilator use in patients with asthma. Subjects suffering from episodic asthma and house dust mite (HDM) allergy usually have a normal lung function testing at rest and show a decrease in lung function when they are exposed to HDM. Bronchial allergen provocation models are well established in asthma research and allow the evaluation of anti-allergic and anti-asthmatic agents in relatively small sample sizes. In a previous study the investigators could show, that LCPUVAs could reduce exhaled NO after repeated BAP with HDM.

In this study the investigators will investigate the protective effect of LCPUVAs in a repeated BAP model. Clinical symptoms (nasal and bronchial), exhaled NO, decrease in lung function the early asthmatic reaction (EAR), the late asthmatic reaction (LAR) and blood parameters (Triglyceride and Cholesterin and mircro RNAs) will be measured before and after LCPUVA supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent

  * Patients: aged ≥18 and 45 years
  * known allergen induced asthma and HDM-Allergy
  * basic lung function FVC ≥ 80%, FEV1 ≥ 75%
  * decrease in FEV1 after BAP ≥ 20%
  * 30% increase of NO after BAP

Exclusion Criteria:

* lung function Forced vital capacity (FVC) <80% and Forced expiratory volume in 1 second (FEV1) <75%
* chronic diseases or infections (e.g. HIV, Tbc)
* pregnancy
* systemic corticosteroid-treatment
* inhalative corticosteroid therapy or leukotriene antagonists
* alcohol, substance or drug abuse
* current smokers
* inability to capture extend and consequences of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Decrase of exhaled NO (eNO) after BAP | 4 weeks
  After BAP with HDM the decrease of eNO will be compared between placebo and active comparator. A relevant decrease is defined as a drop of 30% of exhaled NO.

SECONDARY OUTCOMES:
Absolute levels eNO | 4 weeks
  Comparison of absolute levels eNO (ppb)at end of treatment between groups
Magnitude of EAR | 4 weeks
  Comparison of EAR (maximum decrease of FEV1) at end of treatment between groups
Magnitude of LAR | 4 weeks
  Comparison of LAR (maximum decrease of FEV1 in %) at end of treatment between groups
FEV1 after BAP | 4 weeks
  Comparison of FEV1 Levels 24 hours after BAP between groups
Comparison of methacholin levels | 4 weeks
  Comparison of methacholin (mg) Levels 24 hours after BAP between groups
Asthma control test (ACT) | 4 weeks
  Comparison of ACT score between Groups at end of treatment
Cumulative Salbutamol use | 4 days
  Cumulative Salbutamol use in the last 4 days of treatment during repetitive BAP between groups
Lebel symptom score | 4 weeks
  Comparison of Lebel symptom score after nasal provocation test (NPT), before and after supplementation between groups. A lebel score of 0-4 is negative, a lebel score >5 positive, the maximum result is 12.
Peak nasal expiratory flow | 4 weeks
  Comparison of peak nasal expiratory flow (PNIF) after NPT between groups
Visual analog scala (VAS)-score after NPT | 4 weeks
  Comparison of VAS (mm) after NPT between groups
Visual analog scala (VAS)-score for nasal symptoms | 5 days
  Comparison of cumulative VAS-score for 4 nasal symptoms (Total mm each symptom) in the last 5 days of treatment during repetitive BAP between groups

OTHER OUTCOMES:
Levels of LCPUFA | 4 weeks
  Levels of LCPUFA will be measured before and after Supplementation between groups
Levels of triglyceride and cholesterin | 4 weeks
  Levels of triglyceride and cholesterin will be measured before and after supplementation between groups
Levels of eosinophils | 4 weeks
  Levels of eosinophils will be measured after supplementation and 24 hours after BAP between groups
micro RNAs | 4 weeks
  Levels of micro RNAs will be measured before supplementation and before and 24 hours after BAP between groups

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Professor, Principal Investigator — Klinik für Kinder- und Jugendmedizin Universitätsklinikum
Locations (1):
- Klinik für Kinder- und Jugendmedizin Universitätsklinikum, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be provided of the investigated cohort
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After end of study anticipated June 2020
Access Criteria: The data will be available after the end of study and successful publication of the results (anticipated June 2021 for 10 years